CLINICAL TRIAL: NCT03062059
Title: The Effectiveness and Safety of Intravesical Gemcitabine Instillation During Operation to Prevent Intravesical Recurrence After Radical Nephroureterectomy in Upper Urinary Tract Urothelial Carcinoma: Prospective, Phase II Study
Brief Title: The Effectiveness and Safety of Intravesical Gemcitabine Instillation to Prevent Intravesical Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Seoul National University Hospital (Other); Korea University Anam Hospital (Other); Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, Ho Kyung Seo, Primary Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InstiGem
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Fluid Therapy; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline (Placebo Comparator): Intravesical 52.6ml normal saline instillation during radical nephroureterectomy followed by normal saline bladder irrigation
  Interventions: Other: Normal saline
- Gemcitabine (Experimental): Intravesical 2000mg/52.6ml gemcitabine instillation during radical nephroureterectomy followed by normal saline bladder irrigation
  Interventions: Drug: Intravesical 2000mg/52.6ml gemcitabine instillation

INTERVENTIONS:
Drug: Intravesical 2000mg/52.6ml gemcitabine instillation — Intravesical 2000mg/52.6ml gemcitabine instillation during operation to prevent intravesical recurrence after radical nephroureterectomy in upper urinary tract urothelial carcinoma
  Other Names: Gem Tan inj (liquid)
  Arms: Gemcitabine
Other: Normal saline — Intravesical 52.6ml normal saline instillation after radical nephroureterectomy in upper urinary tract urothelial carcinoma
  Arms: Normal saline

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of intravesical gemcitabine instillation during operation to prevent intravesical recurrence after radical nephroureterectomy in upper urinary tract urothelial carcinoma.

DETAILED DESCRIPTION:
Study Design: Intervention Model: Single Group Assignment

Masking: Open Label

Primary Outcome Measures:

Two year recurrence-free survival in intravesical 2000mg/52.6ml gemcitabine instillation group and control group.

Secondary Outcome Measures:

Time to recurrence in intravesical 2000mg/52.6ml gemcitabine instillation group and control group.

Overall survival in intravesical 2000mg/52.6ml gemcitabine instillation group and control group.

Safety of intravesical 2000mg/52.6ml gemcitabine instillation.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who will undergo nephroureterectomy due to ureter or renal pelvis urothelial carcinoma
* Male or female aged 18 or over 18 years and not more than 85 years who were diagnosed as upper urinary tract urothelial carcinoma
* Normal bone marrow function: Hemoglobin >10 g/dL, ANC >1,500/mm3, platelet count>100,000/mm3
* Normal bladder volume and function
* Normal liver function:
* Bilirubin ≤ 1.5 times of upper normal limit
* AST/ALT ≤ 1.8 times of upper normal limit
* Alkaline phosphatase ≤ 1.8 times of upper normal limit
* Subjects who voluntarily decided to participate and signed the written informed consent

Exclusion Criteria:

* Concomitant bladder cancer
* Subjects who underwent any treatment due to bladder cancer within 3 years
* Prior hypersensitivity reaction history to gemcitabine
* Neurogenic bladder
* Subjects who underwent chemotherapy due to any cancer within 6 months
* Subjects who underwent neoadjuvant chemotherapy due to ureter or renal pelvis urothelial carcinoma
* Hypersensitivity to gemcitabine or component of gemcitabine
* In case of co-administration of gemcitabine and cisplatin in severe renal failure patients
* Moderate to severe liver dysfunction or renal dysfunction (Glomerular filtration rate < 30 mL/min)
* Severe bone marrow suppression
* Severe infection
* Female who are pregnant or has a possibility of pregnancy
* Nursing female
* Interstitial pneumonia or pulmonary fibrosis which is evident on chest x-ray and symptomatic
* Subjects who are undergoing radiotherapy on chest

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Two year recurrence-free survival in intravesical 2000mg/52.6ml gemcitabine instillation group and control group. The recurrence will be assessed by CT scan and cystoscopic exam. | Two years
  Analysis of recurrence status at 2 years from intravesical instillation of 2000mg/52.6ml gemcitabine

SECONDARY OUTCOMES:
Time to recurrence in intravesical 2000mg/52.6ml gemcitabine instillation group and control group. The recurrence will be assessed by CT scan and cystoscopic exam. | six years
  Analysis of time from starting intravesical instillation of 2000mg/52.6ml gemcitabine to recurrence
Overall survival in intravesical 2000mg/52.6ml gemcitabine instillation group and control group. | six years
  Analysis of survival status due to any cause at six years from intravesical instillation of 2000mg/52.6ml gemcitabine
CT cystography finding at one week after surgery. | one week
  Evaluation of leakage at CT cystography at one week from intravesical instillation of 2000mg/52.6ml gemcitabine
International Prostate Symptom Score questionnaire at one week after surgery. | one week
  Evaluation of survey with International Prostate Symptom Score questionnaire a one week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Seok Ho Kang, M.D., Principal Investigator — Korea universitiy
Locations (5):
- South Korea (5):
  - National Cancer Center, Goyang
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No